CLINICAL TRIAL: NCT03757247
Title: Prevalence of Constitutional Mismatch-repair Deficiency Among Suspected Neurofibromatosis Type 1/Legius Syndrome Children Without a Malignancy and Without a NF1 or SPRED1 Mutation
Acronym: CMMRD in NF1
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Other Study IDs: CMMRD_2018
Record Dates: First submitted 2018-11-26; First posted 2018-11-28 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Neurofibromatosis Type 1
MeSH Terms: conditions — Neurofibromatosis 1

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We will analyze at least 670 archived gDNA and cDNA samples of suspected NF1 patients. To avoid generating data for individual patients, we will analyze only fully anonymized samples. However, to get some overall information on the phenotype of the CMMRD patients which will be identified in this study, we will form clinical subgroups within the total cohort.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Frequency of constitutional mismatch-repair deficiency among suspected neurofibromatosis type 1 patients without a NF1 mutation Constitutional mismatch repair deficiency (CMMRD) is a rare inherited condition. Individuals with CMMRD have an extraordinarily high risk to develop a malignant tumor in childhood or adolescence. Nearly all known CMMRD patients developed a malignancy within the first three decades of life and most often in (early) childhood. Since early cancer detection improves the chances to survive, these patients should be included from early childhood on in intensive cancer surveillance protocols. Typically patients are diagnosed with CMMRD only when they develop their first malignant tumor.

Many children with CMMRD show already before the onset of the first malignant tumor clinical signs that may serve as a signpost of this severe condition. Often CMMRD patient show skin patches of milk coffee-like color, termed café au lait maculae (CALM), which are very typical for a different inherited condition named neurofibromatosis type 1 (NF1). NF1, which is much more frequent than CMMRD, also leads to tumor development. But NF1 tumors are usually benign and NF1 children need different, less rigorous, tumor surveillance programs than CMMRD patients. A child with >5 CALM is suspected of having NF1. However, if this diagnosis cannot be confirmed by identification of the causative genetic alteration (NF1-mutation), CMMRD is one possible, but presumably rare, alternative (= differential) diagnosis. Therefore, human geneticists and pediatricians discuss internationally, whether these children should be tested for CMMRD. Diagnosing CMMRD in this situation would allow offering appropriate cancer surveillance protocols to these patients before they develop their first malignant tumor. However, CMMRD testing in this situation may also cause difficulties. Genetic testing may for instance render an ambiguous result, which can neither confirm nor rule out CMMRD. Such a result would create great uncertainty of the appropriate management of the patient. It would be not clear whether intensive cancer surveillance, that may be very stressful for the patient and the family, should be applied or not. Such potential disadvantages of (with respect to tumor development) predictive CMMRD testing argue more against testing when the chances to identify CMMRD in a patient and consequently achieving a benefit for the patient are low. But currently the frequency of CMMRD patients among suspected NF1 patients without a causative NF1 mutation is unknown.

It is the aim of this project to get a reliable estimation on the frequency of the differential diagnosis CMMRD in children with NF1 signs in whom the diagnosis NF1 cannot be confirmed. This information is needed to evaluate and weight the benefits and potential disadvantage of CMMRD testing in these children. To know this frequency is also important for appropriate genetic counseling of at risk children and their parents.

ELIGIBILITY:
Inclusion Criteria:

1. Since CALM or CALM-like pigmentation alterations are the most prevalent NF1 sign in CMMRD patients, at least two should be present in the patient. Therefore, we will include any suspected de novo (=non-familial = NF1 signs absent in parents) NF1 patient who falls into one of three clinical groups:

   1. >5 CALM with or without skinfold freckling and no other NIH NF1 criterion,
   2. >5 CALM with or without skinfold freckling and one or more other NIH NF1 criteria,
   3. 2-5 CALM and one or more NIH NF1 criteria other than CALM.
2. The patient's age must be below 17 years, since the vast majority of CMMRD cases will have developed a tumor by this age. However, overall we aim that the large majority of patients is below the age of 10 years which is the mean age of tumor onset in CMMRD patients.
3. A causative NF1 or SPRED1 mutation must be largely excluded by mutation analysis protocols that reach highest mutation detection rates in bona fide NF1 patients (i.e. familial cases who fulfill NIH criteria)* and sufficient amounts of gDNA and cDNA must be available for subsequent massive-parallel sequencing-based mutation analysis which potentially needs to be complemented with RNA-based techniques (cDNA) particularly for the notoriously difficult PMS2 gene.

Exclusion Criteria:

-

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 670 archived gDNA and cDNA samples of suspectef NF1 patients.
Sampling Method: Probability Sample
Enrollment: 670 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Diagnosis CMMRD | day1
  yes/no